CLINICAL TRIAL: NCT07166588
Title: Convergence Research Platform for the Precision Medicine in the Treatment of Inflammatory Bowel Disease
Brief Title: Research for the Precision Medicine in the Treatment of Inflammatory Bowel Disease
Acronym: PREDICT
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeongJoon Koh, Professor, Seoul National University Hospital
Other Study IDs: 2012-115-1183
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); IBD (Inflammatory Bowel Disease)
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Crohn Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 72 Months
Biospecimen Retention: Samples Without DNA — feces, blood, tissue, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to establish an integrated cohort of patients with inflammatory bowel disease (IBD) from Seoul National University Hospital, Seoul National University Boramae Medical Center, and Seoul National University Bundang Hospital. Through this cohort, we seek to develop a prognostic prediction model for IBD patients and a predictive model for therapeutic responses to biologic agents and small molecule therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10 years or older who have been newly diagnosed with inflammatory bowel disease or are under follow-up monitoring.

Exclusion Criteria:

* Patients diagnosed with cancer or with a history of cancer treatment.
* Participation may be restricted at the discretion of the medical team.
* Infants and young children under the age of 10.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with inflammatory bowel disease, including Crohn's disease and ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction model in the patients with inflammatory bowel disease for treatment response | From enrollment to the end of treatment at 12 weeks
  Development of a prognostic prediction model for patients with inflammatory bowel disease and a predictive model for therapeutic response to biologic agents and small molecule therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea